CLINICAL TRIAL: NCT04412798
Title: Impact of Orange Juice During Breakfast on Glycaemic Control in Individuals With Type 2 Diabetes Mellitus
Brief Title: Orange Juice and Glycaemic Control in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Hochschule Geisenheim University (Unknown)
Responsible Party: Principal Investigator, Dominique Hansen, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Orange -Juice-001
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Other): orange juice concentrate
  Interventions: Other: orange juice concentrate
- Group 2 (Other): Sugar-sweetened orange-flavoured beverage
  Interventions: Other: Sugar-sweetened orange-flavoured beverage
- Group 3 (Other): Whole orange juice with skin removed
  Interventions: Other: Whole orange juice with skin removed

INTERVENTIONS:
Other: orange juice concentrate — 250mL of 100% orange juice made from concentrate
  Arms: group 1
Other: Sugar-sweetened orange-flavoured beverage — Sugar-sweetened orange-flavoured beverage, energy-matched to the orange juice condition
  Arms: Group 2
Other: Whole orange juice with skin removed — Whole orange pieces with skin removed, energy-matched to the orange juice condition
  Arms: Group 3

SUMMARY:
The evidence on the consumption of 100% orange juice in people with type 2 diabetes is highly variable and largely out-of-date, with a few studies reporting acute negative glycaemic effects when 100% orange juice is drunk with or without a meal. The aim of the project is to study the impact of the intake of a single serving of 100% orange juice on glycaemic control in male patients with pre-existing type 2 diabetes mellitus. In addition, immunological parameters and Alzheimer disease related biomarkers will be assessed to examine the chronic inflammatory state of these patients

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: individuals (aged 25-75 years) with up to 8 years of T2DM, according to ADA criteria (Two-hour plasma glucose ≥200 mg/dL (11.1 mmol/L) during OGTT. The test should be performed as described by the WHO, using a glucose load containing the equivalent of 75-g anhydrous glucose dissolved in water; or HbA1c > ≥6.5% (48 mmol/mol)).

Exclusion Criteria:

* pregnancy,
* participants on exogenous insulin therapy,
* HbA1c >8.5%,
* BMI <22 or >35 kg/m²,
* regular smokers (>1 cigarette per day),
* participants with established cardiovascular disease,
* neurological disease,
* cancer,
* renal disease.
* Participants who are unwilling to consume any of the standard foods/drinks

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Glycaemic responses venous blood | baseline
  Venous blood samples collected to examine systemic glycemia (venous blood glucose concentration (mg/dL)) before, during and after a breakfast (differing in supplemented juice composition) for up to 5 hours postprandial.
Glycaemic responses venous blood | Day 5
  Venous blood samples collected to examine systemic glycemia (venous blood glucose concentration (mg/dL)) before, during and after a breakfast (differing in supplemented juice composition) for up to 5 hours postprandial.
Glycaemic responses venous blood | Day 10
  Venous blood samples collected to examine systemic glycemia (venous blood glucose concentration (mg/dL)) before, during and after a breakfast (differing in supplemented juice composition) for up to 5 hours postprandial.
Insulin responses | Baseline
  Venous blood samples collected to examine systemic insulinemia (venous blood insulin concentration (pmol/L)) before, during and after a breakfast (differing in supplemented juice composition) for up to 5 hours postprandial.
Insulin responses | Day 5
  Venous blood samples collected to examine systemic insulinemia (venous blood insulin concentration (pmol/L)) before, during and after a breakfast (differing in supplemented juice composition) for up to 5 hours postprandial.
Insulin responses | Day 10
  Venous blood samples collected to examine systemic insulinemia (venous blood insulin concentration (pmol/L)) before, during and after a breakfast (differing in supplemented juice composition) for up to 5 hours postprandial.
Capillary glycaemic responses | Baseline
  Capillary blood samples collected to examine glycemia before, during and after a breakfast (differing in supplemented juice composition) for up to 5 hours postprandial.
Capillary glycaemic responses | Day 5
  Capillary blood samples collected to examine glycemia before, during and after a breakfast (differing in supplemented juice composition) for up to 5 hours postprandial.
Capillary glycaemic responses | Day 10
  Capillary blood samples collected to examine glycemia before, during and after a breakfast (differing in supplemented juice composition) for up to 5 hours postprandial.

SECONDARY OUTCOMES:
Glycated haemoglobin measure | Baseline
  Measured on a single blood sample to characterize patients' overall glycaemic contro
Flow cytometry | Baseline
  Fasting venous blood samples collected to examine Peripheral blood mononuclear cells (flow cytometry) to measure immunological parameters
Alzheimer disease related biomarkers | Baseline
  Blood samples will be collected every 30 min for 5 hours to examine Alzheimer disease relevant biomarkers (Abeta42, Abeta40, Tau, p-Tau, neuroinflammatory markers and other)
BMI | Baseline
  body weight/height (to determine BMI)
Waist/hip circumference (Body composition) | Baseline
  Waist/hip circumference
Systolic/diastolic blood pressure | Baseline
  Systolic/diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hansen, prof. dr., Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Belgium